CLINICAL TRIAL: NCT03028168
Title: Yôga and Breathing Techniques Training in Patients With Heart Failure and Preserved Ejection Fraction: Study Protocol for a Randomized Clinical Trial
Brief Title: Yôga and Breathing Techniques Training in Patients With Heart Failure and Preserved Ejection Fraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 110069
Record Dates: First submitted 2017-01-16; First posted 2017-01-23 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Cardiovascular Diseases; Heart Failure; Heart Failure, Diastolic
Keywords: Yôga; Breathing Techniques; Heart Failure and Preserved Ejection Fraction
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure; Heart Failure, Diastolic | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention Yôga (Experimental): Active protocol with yôga body movements performed along with respiratory vigorous, without contentions. Two sessions per week, with 45 minutes duration.
  Interventions: Other: Yôga
- Intervention breathing technique (Experimental): Passive protocol, seated patient, no significant body movements. Breathing technique, with alternate nostril breathing combined to inspiratory and expiratory retentions.Two sessions per week, with 45 minutes duration
  Interventions: Other: Breathing technique
- Control group (Experimental): Control group (standard pharmacological treatment). Patients will be oriented to keep their pharmacological routine and daily activities, with no structured exercises. They will have to return to the hospital for post-testing after 8 weeks from randomization.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Yôga — Intervention observing respiratory frequency (RF) of 15- 20 respiratory cycles per minute (rcpm). A standardized 7-minute final relaxation .
  Arms: Intervention Yôga
Other: Breathing technique — Intervention uses diaphragmatic breathing, observing slow respiratory frequency, between 5-8 rcpm. A standardized 7-minute final relaxation.
  Arms: Intervention breathing technique
Other: Control group — Patients will be oriented to keep their pharmacological routine and daily activities, with no structured exercises. They will have to return to the hospital for post-testing after 8 weeks from randomization
  Arms: Control group

SUMMARY:
Current therapies for heart failure (HF) bring together strategies to improve quality of life and exercise tolerance, as well as to reduce morbidity and mortality. Some HF patients present changes in the musculoskeletal system and inspiratory muscle weakness, which may be restored by inspiratory muscle training, thus increasing respiratory muscle strength and endurance, maximum oxygen consumption (VO2), functional capacity, respiratory responses to exercise, and quality of life. Yoga therapies have been shown to improve quality of life, inflammatory markers, and VO2 peak in HF patients, mostly with reduced ejection fraction (HFrEF). However, the effect of different yoga breathing techniques in patients with HF with preserved ejection fraction (HFpEF) has yet to be assessed.

DETAILED DESCRIPTION:
Yôga techniques without breathing control have shown to improve oxygen consumption in patients with HF, mostly HFrEF. However, almost half of HF patients present with HFpEF, and less studies have been performed in those patients. It has been recently demonstrated that HFpEF induces significant molecular, mitochondrial, histological, and functional alterations in the diaphragm and soleus, which were attenuated by exercise training . In cardiac disease and aging, several authors have shown a significant reduction in heart rate variability (HRV) in the frequency ranges associated with breathing, by using spectral analysis of heart rate (HR) and respiration.Therefore, the present randomized clinical trial (RCT) will be conducted in order to test the hypothesis that an program of yôga and specific breathing techniques with different ventilatory rhythms could be associated with improvement in inspiratory muscle responses, functional capacity, oxygen uptake efficiency slope (OUES), circulatory power, oscillatory ventilation, kinetics of oxygen consumption in the recovery period, distinct features of the autonomic nervous system, natriuretic peptides, echocardiographic measurements, and quality of life (QoL) in patients with HFpEF, with and without inspiratory muscle weakness (IMW).Therefore, the present randomized clinical trial (RCT) will be conducted in order to test the hypothesis that an 8-week program of yôga and specific breathing techniques with different ventilatory rhythms could be associated with improvement in inspiratory muscle responses, functional capacity, oxygen uptake efficiency slope (OUES), circulatory power, oscillatory ventilation, kinetics of oxygen consumption in the recovery period, distinct features of the autonomic nervous system, natriuretic peptides, echocardiographic measurements, and quality of life in patients with HFpEF, with and without IMW.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a diagnosis of HFpEF, functional capacity class II and III, who are being treated at a specialized HF clinic will be eligible. HF diagnosis will be established by clinical history (signs and symptoms), echocardiographic findings (left ventricular ejection fraction ≥ 50%) and medical records confirming management for HF.

Exclusion Criteria:

* Pulmonary disease (forced vital capacity<80% of predicted and/or forced expiratory volume in 1 s <70% of predicted, significant mitral or aortic valve diseases, history of exercise-induced asthma, and active smoking or alcoholic.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Maximal inspiratory pressure (PImax) | up to 8 weeks
  Inspiratory muscle strength by measuring maximal inspiratory pressure (PImax)

SECONDARY OUTCOMES:
Peak oxygen uptake (peak VO2) | Baseline and 8 weeks
  Peak VO2 will be considered the highest value of VO2 calculated in a 20-second-period during cardiopulmonary exercise testing (CPET)
Vagal activity: heart rate variability- HRV | Baseline and 8 weeks
  Twenty-four-hour ECG recordings will be obtained with a light digital recorder for to available of heart rate variability (HRV).
Functional capacity through the 6-minute walk test (6MWD) | Baseline and 8 weeks
  The maximum distance walked in 6 minutes of walking (6MWD).The distance traveled in the time of 6 minutes will be considered according to the predicted for gender and age of the patient.
Quality of life Minnesota scores | Baseline and 8 weeks
  Quality of life Minnesota scores as a specific inventory for patients with Heart Failure.
N-terminal pro-brain natriuretic (NT-proBNP) | Baseline and 8 weeks
  NT-proBNP test: N-terminal precursor of natriuretic peptide type B (Brain), clinical specimen by serum, sandwich-type electrochemiluminescence analysis method (COBAS E601-ROCHE).
Echocardiographic - Ejection Fraction | Baseline and 8 weeks
  Teichholz method: ejection fraction - study Inclusion criteria: EF≥ 50% . Establish a diagnostic measure of HF by confirming preserved ejection fraction and compare this measure at the end of the study.

OTHER OUTCOMES:
Other pulmonary functions - Inspiratory muscle force | Baseline and 8 weeks
  Additionally, for the determination of inspiratory muscle force, an incremental test will be used in which patients will breathe continuously through a mouthpiece connected to a measure device. The patients will use an initial load of 50% of PImax, and increments of 10% of PImax will be added every 3 min until the patient is unable to continue breathing.
Oher pulmonary functions - Inspiratory muscle endurance | Baseline and 8 weeks
  Additionally, for the determination of inspiratory muscle endurance, an incremental test will be used in which patients will breathe continuously through a mouthpiece connected to a measure device. The protocol, subjects will breathe against a constant inspiratory submaximal load equivalent to 80% of the greatest inspiratory pressure and the time elapsed to task failure will be defined as the inspiratory endurance time.

CONTACTS AND LOCATIONS:
Overall Officials: Andréia Biolo, MD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (2):
- Brazil (2):
  - Hospital ULBRA - Mãe de Deus, Canoas, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lopes CP, Danzmann LC, Umpierre D, Moraes RS, Soares DS, Leitao SAT, Filho ASC, Depaoli F, Guimaraes LP, Chiappa G, Vieira PJC, Ribeiro JP, Biolo A. YOGA AND BREATHING TRAINING IN PATIENTS WITH HEART FAILURE AND PRESERVED EJECTION FRACTION: A RANDOMIZED CLINICAL TRIAL. medRxiv [Preprint]. 2025 Sep 5:2025.09.03.25335058. doi: 10.1101/2025.09.03.25335058. PMID 40950502
- [Derived] Lopes CP, Danzmann LC, Moraes RS, Vieira PJC, Meurer FF, Soares DS, Chiappa G, Guimaraes LSP, Leitao SAT, Ribeiro JP, Biolo A. Yoga and breathing technique training in patients with heart failure and preserved ejection fraction: study protocol for a randomized clinical trial. Trials. 2018 Jul 28;19(1):405. doi: 10.1186/s13063-018-2802-5. PMID 30055633